CLINICAL TRIAL: NCT06572371
Title: A Prospective Randomized Study Comparing Open Versus Laparoscopic Dismembered Pyeloplasty Among Adult Patients With Primary Pelvi-Ureteric Junction Obstruction
Brief Title: Open Versus Laparoscopic Dismembered Pyeloplasty Among Adult Patients With Primary Pelvi-Ureteric Junction Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mina Soliman Messiha Georgy, Resident of Urology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36133/12/22
Record Dates: First submitted 2024-08-22; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Open; Laparoscopic; Dismembered Pyeloplasty; Primary Pelvi-Ureteric Junction; Obstruction
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic pyeloplasty (Experimental): Patients underwent laparoscopic pyeloplasty.
  Interventions: Procedure: Laparoscopic pyeloplasty
- Open pyeloplasty (Active Comparator): Patients underwent open pyeloplasty.
  Interventions: Procedure: Open pyeloplasty

INTERVENTIONS:
Procedure: Laparoscopic pyeloplasty — The first trocar was inserted under vision through the same supraumbilical incision and the intraperitoneal cavity was inspected The second 5 mm trocar was placed in the midclavicular line 2 inches below the costal margin. The third 10 mm trocar was placed lateral to the rectus muscle at the level of the anterior superior iliac spine. In right-sided pyeloplasty, a fourth trocar was inserted below the xiphistemum for liver retraction. Incision of the line of Toldt and mobilization of the colon was the first step of the transperitoneal approach. A 4/0 polysorbe stay suture was taken in the lateral aspect of the ureter distal to uretero-pelvic junction obstruction to identify the correct orientation after dismembering the ureter. A full thickness anastomosis was started from the angle of V shape spatulation to the lower pole of the renal pelvis.
  Arms: Laparoscopic pyeloplasty
Procedure: Open pyeloplasty — A flank incision with the patient in lateral position was undertaken in open pyeloplasty. After accessing the retro- peritoneum, the ureter was identified and traced cranially till the PUJ segment.
  Traction sutures was placed on the renal pelvis followed by excision of the narrowing segment. The ureter was spatulated by approximately 2 cm and a reduction pyeloplasty was performed, where necessary. Anastomosis was undertaken using vicryl 4-0 sutures. The primary anastomotic site was sutured in interrupted fashion followed by a continuous running suture of the posterior wall. Next, antegrade DJ stenting was performed and the anterior wall was anastomosed. After haemostatic control a 22 Fr drain was placed in the surgical bed.
  Arms: Open pyeloplasty

SUMMARY:
To prospectively compare the perioperative, morphological and functional outcomes on short and medium term between laparoscopic (LP) and open pyeloplasty (OP) patients.

DETAILED DESCRIPTION:
Pelvi-ureteric junction obstruction (PUJO) is defined as a functionally significant impairment of the flow of urine from the kidney's renal pelvis into the proximal ureter.

Open pyeloplasty (OP) has been the gold standard for PUJO repair since the first successful reconstruction of an obstructed PUJO was accomplished in 1892, and achieves success rates exceeding 90%.

Various open surgical techniques have been described based on the cause, location, and length of the PUJO. The most popular repair is the Anderson-Hynes dismembered pyeloplasty, which has universal application and is accepted as the gold standard of treatment.

Now, Laparoscopic dismembered pyeloplasty represents a minimally invasive alternative of gold standard open Anderson- Hynes technique that has a comparable successful outcome with open pyeloplasty while avoiding its co-morbidities. It is also better than endopylotomy as it deals effectively with the crossing vessel

ELIGIBILITY:
Inclusion Criteria:

All adult patients (above 18 years old) with primary pelvi-ureteric junction obstruction indicated for active intervention as

* Symptoms such as recurrent flank pain, recurrent urinary tract infection and rarely hypertension.
* Breakthrough urinary tract infections while on prophylactic antibiotics.
* Increasing renal antero-posterior diameter, or decreasing renal parenchymal thickness by ultrasound.
* Low or decreasing differential renal function, but above 10%.

Exclusion Criteria:

* Patients having poor ipsilateral renal function < 10%.
* Patients with previous pelvi-ureteric junction obstruction repair.
* Associated renal stones.
* Patients unfit for surgery according to American Society of Anesthesiologists classification.
* Contraindications for laparoscopy as (marked obesity, large ventral hernias, gross coagulopathy, abdominal wall sepsis, vertebral deformities…).
* Pediatric patients.
* Pregnant women.
* Vesicoureteral reflux.
* Congenital renal anomalies as (horse- shoe kidney, pelvic kidney, mal- rotated kidney ...).
* Single functioning kidney.
* Malignancy.
* Refusal of written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Amount of blood loss | Intraoperatively
  Amount of blood loss was recorded.

SECONDARY OUTCOMES:
Etiology of obstruction | Intraoperatively
  Etiology of obstruction such as adynamic segment, crossing vessel, stenotic segment, adhesions, and abnormal gonadal vein were recorded.
Complications | 24 hours postoperatively
  Complications was recorded such as wound complications, loin or abdominal pain, fever, chills and rigor, change of color of urine, dysuria.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data was available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data was available upon a reasonable request from the corresponding author.